CLINICAL TRIAL: NCT03714165
Title: Utility of Alpha Defensin and 16S rRNA Gene in Diagnosis of Prosthetic Joint Infection
Brief Title: Alpha Defensin and 16S rRNA Gene in Diagnosis of PJI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Bakhet, Doctor, Assiut University
Other Study IDs: Diagnosis of PJI
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Prosthetic Joint Infection
Keywords: Alpha defensin; 16S rRNA gene

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Alpha defensin and 16SrRNA gene — Alpha defensin 16S rRNA gene CBC: Complete blood count CRP: C reactive protein ESR: Erythrocyte sedimentation rate Culture and antibiotic sensitivity of synovial fluid
  Other Names: CBC; CRP; ESR; Culture and antibiotic sensitivity of synovial fluid

SUMMARY:
Total joint replacement is considered one of the most successful surgical procedures in the field of orthopedics. Despite this achievement, prosthetic joint infections is still considered a severe complication often leading to catastrophic results and requiring repeated and extensive treatment.

The incidence of PJI (a prosthetic joint infection) varies depending on the joint involved; the rate of arthroplasties becoming infected is as follows: 1.7% of primary and 3.2%of non-primary hip arthroplasties.

The accurate diagnosis of prosthetic joint infection often involves the combination of multiple factors including symptoms, signs, synovial fluid cell count, serum inflammatory markers, and culture.

The sensitivity of synovial fluid culture is only 85%, so a negative culture does not rule out infection. However, the specificity of synovial fluid culture is approximately 95%, and positive cultures often imply the presence of prosthetic joint infection.

The synovial fluid alpha-defensin test is an immunoassay that was specifically developed to aid in the diagnosis of prosthetic joint infection .

The sensitivity and the specificity of the alpha-defensin immunoassay test have been reported to be above 96%.

Molecular diagnostic tests using polymerase chain reaction (PCR) are emerging as a tool for the diagnosis of infections and noninfectious conditions. The application of PCR techniques with primers derived from the highly conserved regions of the bacterial 16S rRNA gene has been useful in the detection of bacterial organisms.

Use of broad-range 16S rRNA gene PCR as a tool for identification of bacteria is possible because the 16S rRNA gene is present in all bacteria .

Aim of the work:

.Determine sensitivity and specificity of alpha defensing and 16S rRNA gene in diagnosis of prosthetic joint infection.

* Detection of antibiotic sensitivity for different organisms isolated from synovial fluid

DETAILED DESCRIPTION:
Total joint replacement is considered one of the most successful surgical procedures in the field of orthopedics, alleviating pain and limitation of movement due to degenerative or traumatic joint damage. Despite this achievement, prosthetic joint infections is still considered a severe complication often leading to catastrophic results and requiring repeated and extensive treatment .

Infection is a major problem in orthopedics leading to implant failure. It is a challenging task to treat orthopedic implant infections that may lead to implant replacement and, in severe cases, may result in amputation and mortality Sources of infectious bacteria include the environment of the operating room, surgical equipment, clothing worn by medical and paramedical staff, resident bacteria on the patient's skin and bacteria already residing in the patient's body Implant-associated infections are the result of bacteria adhesion to an implant surface and subsequent biofilm formation at the implantation site .

Staphylococci account for more than 50% of total prosthetic joint infections. Approximately 20% may be polymicrobial, 15% caused by gram-negative, and about 10% are culture negative .

The incidence of PJI (a prosthetic joint infection) varies depending on the joint involved; the rate of arthroplasties becoming infected is as follows: 1.7% of primary and3.2%of non-primary hip arthroplasties .

A correct and early appropriate therapy if correct and timely microbiological diagnosis of infections is done within 4 weeks, it could be possible to follow a conservative approach on the prosthesis, since microorganisms are not yet organized in biofilms. A delayed diagnosis (>4 weeks) of early and late infections involves the necessity of prosthesis removal due to the production of a structured and mature microbial biofilm . The definition of PJI was recently revised by the International Consensus Group on Periprosthetic Joint Infection

According to PJI Consensus Group, patients should be considered to have a PJI if they meet one of the major criteria or at least three of the minor criteria:

Major criteria are as follows:

1. Two positive periprosthetic cultures with phenotypically identical organisms.
2. A sinus tract communicating with the joint.

Minor criteria are as follows:

1. Elevated serum C reactive protein and erythrocyte sedimentation rate.
2. Elevated synovial fluid white blood cell (WBC) count or ++ change on leukocyte esterase test strip.
3. Elevated synovial fluid polymorph nuclear neutrophil percentage.
4. positive histological analysis of periprosthetic tissue.
5. A single positive culture .

Risk factors:

Different pathologies can increase the risk of prosthesis infections: previous infections, obesity, diabetes mellitus, immunodeficiency, and malnutrition or drugs therapy. The clinical assessment provides more details for the suspicion of infection. During physical examination, the surgeon can find the typical inflammation signs as swelling, redness, pain and loss of function .

the most frequent sign was loss of function (95%), followed by pain (85%) and swelling furthermore only 22% of patients presented fever and 14% had feeling of illness but 19% had fistula as primary sign of infection .

Diagnosis:

The accurate diagnosis of prosthetic joint infection often involves the combination of multiple factors including symptoms, signs, synovial fluid cell count, serum inflammatory markers, and culture .

A culture is an important tool for the diagnosis of prosthetic joint infection. Aspirated joint fluid culture should be sent in multiple sets of culture media.

The sensitivity of synovial fluid culture is only 85%, so a negative culture does not rule out infection. However, the specificity of synovial fluid culture is approximately 95%, and positive cultures often imply the presence of prosthetic joint infection .

Numerous preoperative tests for determination and diagnosis of a failed total hip replacement are available. These tests include hematological screening tests (measurement of the erythrocyte sedimentation rate, and the level of C-reactive protein, white blood-cell count,), aspiration of the hip joint, plain radiography, and radionuclide imaging studies. None of these tests is 100 % reliable and are subject to a variable spectrum of false negative or false positive results. A misdiagnosis has crucial consequences for the treatment and for the patient. In case of a misdiagnosed periprosthetic infection, revision of the prosthesis without appropriate debridement would keep a failed total hip replacement and risk an early failure. On the other hand a wrong assumption about periprosthetic infection caused by a false positive test, the patient has to undergo surgery which would be highly inadequate as a girdle stone operation or a cemented revision .

The diagnosis of PJI is based on the clinical findings of arthritis, an abnormal synovial fluid (SF) analysis, and microbiologic confirmation with a positive SF gram stain or culture There are limitations to cultures which may include the following: a delay of at least 2 days from the time of submission for the recovery of the pathogen on the culture medium, the results can be affected by a small inoculum, fastidious organisms may require specialized microbiologic testing, and prior antibiotics may render the culture negative Thus, there is a need for a rapid, sensitive, and specific method in the diagnosis of PJI.

The synovial fluid alpha-defensin test is an immunoassay that was specifically developed to aid in the diagnosis of prosthetic joint infection PJI .

The simplicity of the alpha-defensin test, combined with its ability to provide a clinical result soon after a preoperative joint aspiration, makes it an attractive tool for diagnosing PJI The alpha-defensin protein is an antimicrobial peptide that is naturally released by neutrophils responding to a pathogen in the synovial fluid. It is therefore very reasonable to question whether this antimicrobial peptide is released in response to all pathogens and also whether the alpha-defensin test can detect PJIs caused by all organisms .

The sensitivity and the specificity of the alpha-defensin immunoassay test have been reported to be above 96% .

Use of broad-range 16S rRNA gene PCR as a tool for identification of bacteria is possible because the 16S rRNA gene is present in all bacteria. The 16S rRNA gene consists of highly conserved nucleotide sequences, interspersed with variable regions that are genus- or species-specific.

Molecular diagnostic tests using polymerase chain reaction (PCR) are emerging as a tool for the diagnosis of infections and noninfectious conditions. The application of PCR techniques with primers derived from the highly conserved regions of the bacterial 16S rRNA gene has been useful in the detection of bacterial organisms.

ELIGIBILITY:
Inclusion Criteria:

- The study will include all patient with prosthetic joint suspected to be infected through clinical manifestation (fever, pain, fistula redness, swelling ,hotness and loss of function) associated with radiological evidence.

Exclusion Criteria:

* Any patient began antibiotic treatment will be excludes from the samples.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted on 90 informed individuals (according to guidelines of ethical committee of faculty of medicine , Assuit University )
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of Alpha defensin in diagnosis of Prosthetic joint infection | 2 days
  value of measuring Alpha defensin by enzyme linked immunosorbent assay (ELISA) in diagnosis of Prosthetic joint infection as a rapid bio marker
Diagnostic value of 16S rRNA gene in diagnosis of Prosthetic joint infection | 2 days
  value of measuring 16S rRNA gene by conventional PCR in diagnosis of Prosthetic joint infection as more accurate test

CONTACTS AND LOCATIONS:
Overall Officials: Osama Bakr Sedek, MD, Principal Investigator — Assuit Univeristy; Dalia Tarik Kamal, MD, Study Chair — Assuit Univeristy; Amal Mohammed Hosney, MD, Study Chair — Assuit Univeristy; Ayat Bakhet Mostafa, Dr, Study Director — Assuit Univeristy
Locations (1):
- Ayat Bakhet Mostafa, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slullitel PA, Onativia JI, Buttaro MA, Sanchez ML, Comba F, Zanotti G, Piccaluga F. State-of-the-art diagnosis and surgical treatment of acute peri-prosthetic joint infection following primary total hip arthroplasty. EFORT Open Rev. 2018 Jul 17;3(7):434-441. doi: 10.1302/2058-5241.3.170032. eCollection 2018 Jul. PMID 30233819
- [Background] Dudareva M, Barrett L, Figtree M, Scarborough M, Watanabe M, Newnham R, Wallis R, Oakley S, Kendrick B, Stubbs D, McNally MA, Bejon P, Atkins BA, Taylor A, Brent AJ. Sonication versus Tissue Sampling for Diagnosis of Prosthetic Joint and Other Orthopedic Device-Related Infections. J Clin Microbiol. 2018 Nov 27;56(12):e00688-18. doi: 10.1128/JCM.00688-18. Print 2018 Dec. PMID 30209185